CLINICAL TRIAL: NCT00415285
Title: Randomized Phase II Trial of Sequential Docetaxel Followed by Capecitabine Versus Concomitant Docetaxel/Capecitabine as in Induction Therapy for Early Stage Breast Cancer
Brief Title: Docetaxel Followed by Capecitabine Versus Concomitant Docetaxel/Capecitabine for Early Stage Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Georgia Center for Oncology Research & Education (Other)
Collaborators: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EU822-03
Record Dates: First submitted 2006-12-20; First posted 2006-12-22 (Estimated); Last update posted 2007-02-13 (Estimated); Status verified 2007-02

CONDITIONS: Breast Neoplasms
Keywords: Breast; Cancer; Early-Stage; Chemotherapy
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — Docetaxel; Capecitabine

INTERVENTIONS:
Drug: Docetaxel
Drug: Capecitabine
Drug: Docetaxel/Capecitabine

SUMMARY:
The purpose of this study is to identify new chemotherapy treatment regimens with better response rates and to find out if the combination of docetaxel and capecitabine can shrink the size of breast tumors and preserve the breast.

DETAILED DESCRIPTION:
The purpose of this study is to identify new chemotherapy treatment regimens with better response rates and to find out if the combination of docetaxel and capecitabine can shrink the size of breast tumors and preserve the breast.

Induction chemotherapy offers the possibility of less surgery and determines tumor sensitivity in vivo. Previous trials have demonstrated that complete pathologic response in the breast at surgery corresponds with improved outcome. Additionally, we will correlate specific molecular markers in the breast tumors before and after chemotherapy, with response to treatment.

Expression of these molecular markets may be used in the future to predict the likelihood of response to chemotherapy given post-operatively.

Approximately 100 patients will participate at Emory Winship Cancer Institute and Emory Crawford W. Long Hospital and Grady Health System in Atlanta, Georgia.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed breast carcinoma.
* Early stage breast cancer (stage 1, 2, 3).
* No evidence of disease outside the breast or chest wall, except ipsilateral axillary lymph nodes.
* 18 years of age or older.
* Final eligibility for a clinical trial is determined by the health professionals conducting the trial.

Exclusion Criteria:

* Prior chemotherapy, hormonal therapy, biologic therapy or radiation therapy for breast cancer.
* Major surgery within 28 days of study entry.
* Evidence of CNS metastases.
* Final eligibility for a clinical trial is determined by the health professionals conducting the trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2006-12

CONTACTS AND LOCATIONS:
Overall Officials: Ruth O'Regan, MD, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Grady Memorial Hospital, Atlanta, Georgia
  - Emory Crawford Long Hospital, Atlanta, Georgia
  - Winship Cancer Institute of Emory University, Atlanta, Georgia

REFERENCES:
- See also: Winship Cancer Institute — http://www.winshipcancerinstitute.org/